CLINICAL TRIAL: NCT06914895
Title: A Phase 3, Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study Evaluating the Efficacy and Safety of Tirzepatide Once Weekly Compared to Placebo in Adult Participants With Type 1 Diabetes and Obesity or Overweight
Brief Title: A Study of Tirzepatide (LY3298176) Compared With Placebo in Adults With Type 1 Diabetes and Obesity or Overweight
Acronym: SURPASS-T1D-1
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 27285; I8F-MC-GPJA (Other: Eli Lilly and Company); 2024-519684-17-00 (EU CTIS Number)
Record Dates: First submitted 2025-04-04; First posted 2025-04-06 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Type 1 Diabetes; Obesity; Overweight
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Obesity; Overweight | interventions — Tirzepatide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Tirzepatide Dose 1 (Experimental): Participants will receive tirzepatide subcutaneously (SC)
  Interventions: Drug: Tirzepatide
- Tirzepatide Dose 2 (Experimental): Participants will receive tirzepatide SC
  Interventions: Drug: Tirzepatide
- Tirzepatide Dose 3 (Experimental): Participants will receive tirzepatide SC
  Interventions: Drug: Tirzepatide
- Tirzepatide Dose 4 (Experimental): Participants will receive tirzepatide SC
  Interventions: Drug: Tirzepatide
- Placebo (Placebo Comparator): Participants will receive placebo SC
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tirzepatide — Administered SC
  Other Names: LY3298176
  Arms: Tirzepatide Dose 1; Tirzepatide Dose 2; Tirzepatide Dose 3; Tirzepatide Dose 4
Drug: Placebo — Administered SC
  Arms: Placebo

SUMMARY:
The main purpose of this study is to find out how well and how safely tirzepatide works in adults who have type 1 diabetes and obesity or overweight. Participation in the study will last about 49 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Have type 1 diabetes and on insulin treatment for at least one year prior to screening
* Have an HbA1c value of 7.0% to 10.5% inclusive, at screening
* Have a body mass index (BMI) of ≥25 kilograms per square meter (kg/m2) at screening
* Are of stable weight for at least 90 days prior to screening and agree to not start an intensive diet or exercise program during the study

Exclusion Criteria:

* Have experienced two or more events requiring hospitalization due to poor glucose control (hyperglycemia or (diabetic ketoacidosis (DKA)) during the period of 180 days prior to screening and until randomization.
* Have experienced one or more events of severe hypoglycemia during the period of 90 days prior to screening and until randomization.
* Are currently receiving or planning to receive treatment for diabetic retinopathy and/or macular edema
* Have had chronic or acute pancreatitis
* Have used any weight loss drugs or alternative remedies, including herbal or nutritional supplements, within 90 days prior to screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 905 (Estimated)
Dates: Start 2025-04-25 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Hemoglobin A1c (HbA1c) | Baseline, Week 40

SECONDARY OUTCOMES:
Percentage of Time Continuous Glucose Monitor (CGM) Glucose Values are Between 70 and 180 milligrams per deciliter (mg/dL) (3.9 and 10.0 millimoles per liter (mmol/L) Inclusive, Per Day | Within 30 days prior to Week 40
Change from Baseline in Body Weight | Baseline, Week 40
Percent Change from Baseline in Body Weight | Baseline, Week 40
Percentage of Participants with ≥5% Body Weight Reduction | Baseline, Week 40
Percentage of Participants with ≥10% Body Weight Reduction | Baseline, Week 40
Percentage of Participants with ≥15% Body Weight Reduction | Baseline, Week 40
Change from Baseline in Waist Circumference | Baseline, Week 40
Change from Baseline in Systolic Blood Pressure (SBP) | Baseline, Week 40
Percent Change from Baseline in Fasting Triglycerides | Baseline, Week 40
Percent Change from Baseline in Fasting Non-High-Density Lipoprotein (non-HDL) Cholesterol | Baseline, Week 40
Percent Change from Baseline in Total Daily Insulin Dose | Baseline, Week 40
Percent Change from Baseline in High-Sensitivity C-Reactive Protein (hsCRP) | Baseline, Week 40
Change from Baseline in EQ-5D-5L | Baseline, Week 40

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 8 AM - 8 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (146):
- United States (31):
  - Sansum Diabetes Research Institute, Santa Barbara, California
  - Care Access - Santa Clarita, Santa Clarita, California
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - Atlanta Diabetes Associates, Atlanta, Georgia
  - Orita Clinical Research, Decatur, Georgia
  - North Georgia Clinical Research, Woodstock, Georgia
  - East-West Medical Research Institute, Honolulu, Hawaii
  - Rocky Mountain Clinical Research, Idaho Falls, Idaho
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Indiana University Health University Hospital, Indianapolis, Indiana
  - Iowa Diabetes and Endocrinology Research Center, West Des Moines, Iowa
  - Endocrine and Metabolic Consultants, Rockville, Maryland
  - HealthPartners Institute dba International Diabetes Center, Minneapolis, Minnesota
  - SKY Integrative Medical Center/SKYCRNG, Ridgeland, Mississippi
  - Boeson Research MSO, Missoula, Montana
  - Palm Research Center Tenaya, Las Vegas, Nevada
  - Palm Research Center Sunset, Las Vegas, Nevada
  - Albany Medical College, Division of Community Endocrinology, Albany, New York
  - Research Foundation of SUNY - University of Buffalo, Buffalo, New York
  - NYC Research, New York, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - Lucas Research, Inc., Morehead City, North Carolina
  - Care Access - Lima, Lima, Ohio
  - Alliance for Multispecialty Research, LLC, Norman, Oklahoma
  - Suburban Research Associates, West Chester, Pennsylvania
  - Texas Diabetes & Endocrinology, P.A., Austin, Texas
  - Velocity Clinical Research, Dallas, Dallas, Texas
  - Tekton Research, LLC., McKinney, Texas
  - Medrasa Clinical Research, Wylie, Texas
  - Eastside Research Associates, Redmond, Washington
  - Rainier Clinical Research Center, Renton, Washington
- Argentina (12):
  - Investigaciones Medicas Imoba Srl, Buenos Aires
  - Centro de Investigaciones Metabólicas (CINME), Buenos Aires
  - CIPREC, Buenos Aires
  - Consultorio de Investigación Clínica EMO SRL, Buenos Aires
  - CENUDIAB, Buenos Aires
  - Instituto de Investigaciones Clínicas Córdoba, Córdoba
  - Centro Medico Privado San Vicente Diabetes, Córdoba
  - Centro de Investigaciones Médicas Mar del Plata, Mar del Plata
  - Instituto Médico Río Cuarto, Río Cuarto
  - Fundacion Estudios Clinicos, Rosario
  - Centro de Diagnóstico y Rehabilitación (CEDIR), Santa Fe
  - Centro de Salud e Investigaciones Médicas, Santa Rosa
- Brazil (10):
  - Centro de Diabetes Curitiba, Curitiba
  - Centro De Diabetes Metabolismo E Endocrinologia, Fortaleza
  - Private Practice - Dr.Miguel N. Hissa, Fortaleza
  - Universidade Federal de Goias, Goiânia
  - CPQuali Pesquisa Clínica, São Paulo
  - CPCLIN, São Paulo
  - IBTED - Tecnologia e Educação em Diabetes, São Paulo
  - CEPIC - Centro Paulista de Investigação Clínica, São Paulo
  - Hospital das Clinicas FMUSP, São Paulo
  - CEDOES, Vitória
- Denmark (5):
  - Esbjerg sygehus, Syddansk Universitetshospital, Esbjerg
  - Steno Diabetes Center - Copenhagen, Herlev
  - Regionshospitalet Gødstrup, Herning
  - Nordsjællands Hospital - Hillerød, Hillerød
  - Sjællands Universitetshospital Køge, Køge
- France (13):
  - Centre Hospitalier Universitaire de Caen - Hôpital Côte de Nacre, Caen
  - Centre Hospitalier Sud Francilien, Corbeil-Essonnes
  - Hôtel-Dieu du Creusot - site Harfleur, Le Creusot
  - Centre du diabète DIAB-eCARE, Lyon
  - Hôpital Européen Marseille, Marseille
  - Hôpital de la Conception, Marseille
  - CHU Montpellier Lapeyronie Hospital, Montpellier
  - Hôpital Nord Guillaume-et-René-Laennec / CHU de Nantes, Nantes
  - Hôpital NOVO, Pontoise
  - CHU Strasbourg-Hautepierre, Strasbourg
  - Centre Hospitalier intercommunal de Toulon La Seyne sur Mer, Toulon
  - CHU Rangueil, Toulouse
  - Groupe Hospitalier Mutualiste Les Portes du Sud, Vénissieux
- Germany (9):
  - Diabetespraxis Mergentheim, Bad Mergentheim
  - Diabetes- und Stoffwechselpraxis Bochum, Bochum
  - InnoDiab Forschung Gmbh, Essen
  - Diabetes Zentrum Wilhelmsburg, Hamburg
  - Klinikum Karlsburg, Karlsburg
  - Universitätsklinikum Leipzig, Leipzig
  - Institut für Diabetesforschung GmbH Münster, Münster
  - RED-Institut GmbH, Oldenburg
  - Arztpraxis Christine Kosch Pirna, Pirna
- Israel (10):
  - Yitzhak Shamir Medical Center, Beer Yaacov
  - Soroka Medical Center, Beersheba
  - Rambam Health Care Campus, Haifa
  - Institute of Diabetes, Technology and Research - Clalit Health, Herzliya
  - Hadassah Medical Center, Jerusalem
  - Schneider Children's Medical Center, Petah Tikva
  - Rabin Medical Center, Petah Tikva
  - Sheba Medical Center, Ramat Gan
  - Diabetes Medical Center, Tel Aviv
  - Sourasky Medical Center, Tel Aviv
- Italy (8):
  - IRCCS - AOU di Bologna, Bologna
  - AOU Renato Dulbecco, Catanzaro
  - Azienda Ospedaliera Universitaria Careggi, Florence
  - Ospedale San Raffaele, Milan
  - University of Naples Federico II, Napoli
  - Azienda Ospedale - Università Padova, Padua
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS - Università Cattolica del Sacro Cuore, Roma
  - Azienda Ospedaliero-Universitaria Città della Salute e della Scienza di Torino, Torino
- Japan (29):
  - The Institute of Medical Science, Asahi Life Foundation, Chūōku
  - Matoba Internal Medicine Clinic, Ebina
  - Clinic Masae Minami, Fukuoka
  - Japanese Red Cross Fukuoka Hospital, Fukuoka
  - Hachioji Diabetes Clinic, Hachioji-shi
  - Takai Internal Medicine Clinic, Kamakura-shi
  - Shiraiwa Medical Clinic, Kashiwara
  - Kasugai Municipal Hospital, Kasugai
  - Kimitsu Chuo Hospital, Kisarazu
  - Yamanashi Prefectural Central Hospital, Kofu
  - Kumamoto Central Hospital - Kumamoto, Kumamoto
  - Jinnouchi Hospital, Kumamoto
  - Kure Medical Center, Kure
  - Mikannohana Clinic, Diabetes, Endocrinology and Metabolism, Matsuyama
  - Kozawa Eye Hospital and Diabetes Center, Mito
  - Heiwadai Hospital, Miyazaki
  - Soleil Chikusa Clinic, Nagoya
  - Tosaki Clinic for Diabetes and Endocrinology, Nagoya
  - Nakakinen clinic, Naka
  - Osaka City General Hospital, Osaka
  - Abe Clinic, Ōita
  - Odori Diabetes, Sapporo
  - Manda Memorial Hospital, Sapporo
  - Shimonoseki Medical Center, Shimonoseki
  - Tomonaga Clinic, Shinjuku
  - Suruga Clinic, Shizuoka
  - Tama Center Clinic Mirai, Tama
  - Noritake Clinic, Ushiku
  - Japanese Red Cross Society - Wakayama Medical Center, Wakayama
- Mexico (9):
  - Enclifar Ensayos Clínicos Farmacológicos Sc, Chihuahua City
  - Unidad de Investigaci�n Cl�nica Cardiometabolica de Occidente, Guadalajara
  - Centro de Investigacion Medica de Occidente, S.C., Guadalajara
  - Unidad de Investigación Clínica y Atención Médica HEPA S.C., Guadalajara
  - Invecordis S.C., Hacienda de Las Palmas
  - CEINV Salud, Monterrey
  - Clínica García Flores SC, Monterrey
  - Consultorio Médico de Endocrinología y Pediatría, Puebla City
  - Medsal Centro Médico, Tampico
- Puerto Rico (2):
  - Advanced Clinical Research, LLC, Bayamón
  - Manati Center for Clinical Research, Manatí
- Spain (8):
  - CHUAC-Complejo Hospitalario Universitario A Coruña, A Coruña
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Complejo Hospitalario Universitario de Ferrol (CHUF)- Hospital Naval, Ferrol
  - Hospital Universitario de Móstoles, Móstoles
  - Hospital Universitario Marqués de Valdecilla, Santander
  - Hospital Universitario Virgen Del Rocio, Seville

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- See also: A Study of Tirzepatide (LY3298176) Compared With Placebo in Adults With Type 1 Diabetes and Obesity or Overweight (SURPASS-T1D-1) — https://trials.lilly.com/en-US/trial/589916